CLINICAL TRIAL: NCT02275845
Title: Metformin vs Control to Prevent Gestational Diabetes Mellitus (GDM) in Women With a High Risk for GDM, an Open Label Randomized Controlled Trial, The Medico-GDM Trial
Brief Title: Medico-GDM Trial - Metformine to Prevent Gestational Diabetes Mellitus
Acronym: Medico-GDM
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Maasstad Hospital (Other)
Responsible Party: Principal Investigator, Wetenschapsbureau, dr. J. van der Linden, Maasstad Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NL48005.101.15; 2014-000446-30 (EudraCT Number)
Record Dates: First submitted 2014-10-23; First posted 2014-10-27 (Estimated); Last update posted 2015-12-28 (Estimated); Status verified 2015-12

CONDITIONS: Gestational Diabetes Mellitus
Keywords: metformin; prevention
MeSH Terms: conditions — Diabetes, Gestational | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- intervention (Experimental): Metformin twice daily 500 mg for the first week, after that twice daily 1000 mg. All the subjects are receiving a diet which contains a 2000 calories/day diet, with an adequate distribution of carbohydrates during the day.
  Interventions: Drug: Metformin; Other: control diet
- control diet (Active Comparator): a diet which contains a 2000 calories/day diet, with an adequate distribution of carbohydrates during the day.
  Interventions: Other: control diet

INTERVENTIONS:
Drug: Metformin — Metformin twice daily 500 mg for the first week, after that twice daily 1000 mg (from 14 weeks pregnancy untill delivery)
  Arms: intervention
Other: control diet — 2000 calories/day diet, with an adequate distribution of carbohydrates during the day

SUMMARY:
Metformin vs Control to prevent gestational diabetes mellitus (GDM) in women with a high risk for GDM, an open label randomized controlled trial' The Medico-GDM trial

DETAILED DESCRIPTION:
Rationale: GDM is a frequent pregnancy complication1 and associated with complications for mother and child.2 At present, the drug of choice for treatment of GDM is Insulin.3 In the last years several studies documented the use of oral blood glucose lowering medication in GDM. Metformin is an accepted alternative for insulin, with comparable glycemic control and neonatal outcomes.4 In studies with women with polycystic ovarian syndrome (PCOS) who received Metformin during pregnancy, the incidence of GDM is less compared to pregnant women with PCOS without Metformin. These studies were however small and there was no adequate control group.5 Our aim is to study the effect of Metformin on the incidence of GDM in women with a high risk for GDM.

Objective: the primary objective is to compare metformin versus no intervention for incidence of GDM in women with a high risk for GDM. The main secondary objective is pregnancy outcome with Metformin, neonatal outcomes and neonatal complications.

Study design: 2 years open label randomized controlled trial, comparing metformin versus control group.

Study population: pregnant women with a high risk of GDM between 18 and 40 years old in the first trimester of pregnancy.

Intervention: the first group receives Metformin twice daily 500 mg for the first week, after that twice daily 1000 mg. The second group receives no intervention. All the subjects are receiving a diet which contains a 2000 calories/day diet, with an adequate distribution of carbohydrates during the day.

Main study parameters/endpoints: the main study parameter is the difference in incidence of GDM between the two groups.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: the subjects will visit our centre for the first time between 12 and 14 weeks of pregnancy, then blood samples will be collected. Further on they will visit our centre at 24 weeks to perform an oral glucose tolerance test (OGTT). Women with GDM in history will perform an OGTT at 16 weeks for the first time. If the OGTT is borderline normal, it will repeated every 4 weeks. This is according to current Dutch guidelines3, without any extra discomfort for study participants. The subjects will visit their own gynaecologist or obstretican for their regular pregnancy controls. Metformin is not officially registered for use in pregnancy. Long term effects for the unborn child are not known. However, previous studies did not found neonatal and pregnancy related complications.

ELIGIBILITY:
Inclusion Criteria:

a subject must meet all of the following criteria:

* high risk (according to ductch national criteria) for gestational diabetes
* aged between 18 and 40 years
* gestational age between 8 and 12 weeks
* and able to communicate and read in Dutch.

Exclusion Criteria:

A potential subject who meets any of the following criteria will be excluded from participation in this study:

* no singleton pregnancy judged by ultrasonography
* diagnosis of diabetes mellitus before the current pregnancy-
* high fasting glucose at first trimester (> 5.3 mmol/l)
* cardiac insufficiency-\
* renal insufficiency (MDRD < 60)
* liver disease
* use of medication other than Paracetamol or vitamins and incompetent women.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 400 (Estimated)
Dates: Start 2014-09; Primary Completion 2016-09 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
incidence of gestational diabetes mellitus in both groups | from 14 weeks pregnancy untill delivery

SECONDARY OUTCOMES:
Maternal outcomes | from 14 weeks pregnancy untill delivery
  Maternal: pregnancy induced hypertension (yes vs no: systolic blood pressure ≥140 mmHg or diastolic blood pressure ≥90 mmHg), weight gain during pregnancy (kg), abnormal glucose daily curve after pregnancy (yes vs no: measurement of blood glucose concentration seven times daily).), insulin therapy required.
Neonatal outcomes | from 14 weeks pregnancy untill delivery
  head circumference (cm), birth weight (g) and height (cm), pH of umbilical-cord.
  Neonatal complications: serious neonatal complications (including: severe birth defects, stillbirth, birth trauma, respiratory distress, admission to neonatal intensive care unit, low 5-minutes Apgar score (< 7) and premature birth (< 37 weeks of gestation)), neonatal hypoglycaemia that requires therapy, need for phototherapy, small for gestational age (birth weight < 2 SD units), birth weight > 90th percentile, birth weight < 10th percentile.

CONTACTS AND LOCATIONS:
Overall Officials: Joke van der Linden, dr., Principal Investigator — Maasstad Hospital
Locations (1):
- Maasstad Ziekenhuis, Rotterdam, Netherlands